CLINICAL TRIAL: NCT07040332
Title: Pathogenesis and Inflammatory Phenotype of Allergic Bronchopulmonary Aspergillosis
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Tongji University School of Medicine (Unknown); Fudan University (Other); Guizhou Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qian Qi, Dr., Qianfoshan Hospital
Other Study IDs: QFS-2025-074
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Allergic Bronchopulmonary Aspergillosis (ABPA)
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- allergic bronchopulmonary aspergillosis
- fungal-sensitized asthma
- control group

INTERVENTIONS:
Other:  — No intervention

SUMMARY:
This study aims to reveal the immune and inflammatory regulatory molecular mechanisms related to the progression of allergic bronchopulmonary aspergillosis (ABPA), and to build a precision typing based on inflammation and identify the biomarkers of typing, and to explore the clinical outcomes of different inflammatory phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for allergic bronchopulmonary aspergillosis.
* Meets the diagnostic criteria for fungal-sensitized asthma.

Exclusion Criteria:

* Human immunodeficiency virus infection.
* Malignant tumor.
* Blood system disease.
* autoimmune system disease.
* History of pulmonary tuberculosis.
* Patients with a history of smoking or still smoking.
* Invasive pulmonary fungal disease.
* Contraindications electronic bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with allergic bronchopulmonary aspergillosis and fungal-sensitized asthma who were treated in several hospitals were included as the study objects, and the relatively normal ones who had no bronchial asthma and no fungal sensitization were matched by gender and age as the control group, and then the cohorts of patients with allergic bronchopulmonary aspergillosis, fungal-sensitized asthma and the control group were established.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Total serum IgE | Up to 12 months

SECONDARY OUTCOMES:
Aspergillus-specific IgE | Up to 12 months
Aspergillus-specific IgG | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No